CLINICAL TRIAL: NCT01314131
Title: Use of Autobiographical and Interest Assessment for a Better Stimulation of Patients in Nursing Home
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association Recherche Méthodologie Evaluation Psychiatrique (Other)
Responsible Party: Pr ROBERT Philippe, Centre Mémoire de Ressources et de Recherche
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ARMEP-01
Record Dates: First submitted 2011-03-11; First posted 2011-03-14 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention group (Experimental)
  Interventions: Behavioral: Stimulation group

INTERVENTIONS:
Behavioral: Stimulation group — Patients living in nursing home can be enrolled in the study by giving their verbal consent. The trial lasts two weeks for each patients and it will be performed in three parts :
  * a cognitive and behaviour assessment : MMSE, BREF, NPI, IA
  * an interest questionnaire for patients. It contains 40 questions about activities.
  * the intervention : patients will be propose 5 activities. 4 of them are activities that patients are interested in. Each activity have to last 15 minutes and the stimulation is measured by a scale named "Observational Measurement of Engagement ".
  Other Names: interest; autobiography

SUMMARY:
The purpose is to evaluate patients' interests (patients in nursing home). Moreover the study aims to evaluate whether an activity for which the patient is interested in, allows a better involvement and stimulation.

DETAILED DESCRIPTION:
Context :

Behavioral and Psychological Symptoms of Dementia (BPSD) arouse researchers' interest because they are frequent manifestations responsible for a large share of the suffering of patients and caregivers. Apathy is the most frequent of them.

Systematic literature reviews on non-pharmacological treatment for BPSD indicates that some technique and more particularly residential care staff training program appear to have promising results, even if the level of evidence of efficacy remains moderate partly because of the paucity of scientific quality research in this area.

The most of them comes from Anglo-Saxon country. In France, the TNM en EHPAD study demonstrated the staff training program efficacy regarding to the management of behavioral positive symptoms such as agitation or aggressiveness compared to a control group

Aims of the study :

The aims of the study is to evaluate the short and medium term effectiveness of staff training program to manage and stimulate patients with a diagnosis of Alzheimer's disease or associated disorders and presenting BPSD of the apathy type and living in nursing homes.

Description :

A Randomized controlled trial (randomization by nursing home) presents as a routine clinical procedure according to the French regulation. Raters and our statistician are unaware and blind to the randomization. The trial takes place in 4 nursing homes.

To be included, patients are older than 65 years with a diagnosis of Alzheimer's disease or associated disorder and present the diagnostic criteria of apathy, within a moderate to severe stage of the disease.

Data are collected at baseline, month 1 and at month 4, namely 3 months after the end of the training programme thanks to the Apathy Inventory Clinician version (AI-C), the Neuropsychiatric Inventory for the staff members (NPI-ES), the AD QOL, an Observation Scale and a qualitative analysis of the official caregiver's knowledge and perception about BPSD especially apathy and their expectations concerning the training program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimer's disease
* MMSE score between 12 and 24
* Patient involved in organized activities in nursing home

Exclusion Criteria:

Patients:

* Who are not able to understand and answer to questions for the study
* < 60 years of age
* Who are not able to sit
* Aphasic

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-09 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the engagement duration for an activity, measured by the OME (Observational Measurement of Engagement) scale. | 10 times during two weeks
  First, a cognitive and behaviour assessment (specially autobiographical memory) is performed to patients.
  Then, the patient is proposed to do 5 activities. 4 of them correpond to activities for which he is interested in (depending on the assessment results). The therapist assesses if the patient is stimulated, by measuring the time for which he is involved in doing the activity (with OME Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ROBERT, PhD, Principal Investigator — Centre Mémoire de Ressources et de Recherche
Locations (1):
- Centre Mémoire de Ressources et de Recherche, Nice, France